CLINICAL TRIAL: NCT02493751
Title: A PHASE 1B, OPEN-LABEL, DOSE-FINDING STUDY TO EVALUATE SAFETY, PHARMACOKINETICS AND PHARMACODYNAMICS OF AVELUMAB (MSB0010718C) IN COMBINATION WITH AXITINIB (AG-013736) IN PATIENTS WITH PREVIOUSLY UNTREATED ADVANCED RENAL CELL CANCER
Brief Title: A Study Of Avelumab In Combination With Axitinib In Advanced Renal Cell Cancer (JAVELIN Renal 100)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Masking: None | Purpose: Treatment
Other Study IDs: B9991002; 2015-001137-25 (EudraCT Number); Javelin Renal 100 (Other: Alias Study Number)
Record Dates: First submitted 2015-07-07; First posted 2015-07-09 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-12

CONDITIONS: Renal Cell Cancer
Keywords: Cancer, renal cell cancer, kidney disease, kidney neoplasms, axitinib
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Kidney Diseases; Kidney Neoplasms | interventions — avelumab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose finding phase and dose expansion phase. (Experimental): To test the maximum tolerated dose of avelumab (MSB0010718C) in combination with axitinib (AG-013736)
  Interventions: Drug: Avelumab (MSB0010718C); Drug: Axitinib (AG-013736)

INTERVENTIONS:
Drug: Avelumab (MSB0010718C) — Avelumab with two dose levels: 10 mg/kg IV and 5 mg/kg IV every two weeks to find the maximum tolerated dose in combination with axitinib and continue treatment in a dose expansion.
Drug: Axitinib (AG-013736) — Axitinib with two dose levels: 5 mg and 3 mg oral BID to find the maximum tolerated dose in combination with avelumab and continue treatment in a dose expansion.

SUMMARY:
This is a Phase 1b, open-label, multi-center, multiple-dose trial designed to estimate the maximum tolerated dose (MTD) and select the recommended phase 2 dose (RP2D) of avelumab (MSB0010718C) in combination with axitinib (AG-013736). Once the MTD of avelumab administered in combination with axitinib is estimated (dose finding portion), the dose expansion phase will be opened to further characterize the combination in term of safety profile, anti tumor activity, pharmacokinetics, pharmacodynamics and biomarker modulation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced RCC with clear cell component
* Primary tumor resected
* Availability of a recent formalin-fixed, paraffin-embedded (FFPE) tumor tissue block from a de novo tumor biopsy during screening (biopsied tumor lesion should not be a RECIST target lesion). Alternatively, a recently obtained archival FFPE tumor tissue block (not cut slides) from a primary or metastatic tumor resection or biopsy can be provided if the following criteria are met: 1) the biopsy or resection was performed within 1 year of enrollment AND 2) the patient has not received any intervening systemic anti-cancer treatment from the time the tissue was obtained and enrollment onto the current study. If an FFPE tissue block cannot be provided as per documented regulations,, 15 unstained slides (10 minimum) will be acceptable.
* Availability of an archival FFPE tumor tissue block from primary diagnosis specimen (if available and not provided per above). If an FFPE tissue block cannot be provided, 15 unstained slides (10 minimum) will be acceptable
* At least one measureable lesion as defined by RECIST version 1.1 that has not been previously irradiated.
* Age ≥18 years (≥ 20 years in Japan).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate bone marrow function, renal and liver functions

Exclusion Criteria:

* Prior systemic therapy directed at advanced RCC.
* Prior adjuvant or neoadjuvant therapy for RCC if disease progression or relapse has occurred during or within 12 months after the last dose of treatment
* Prior immunotherapy with IL-2, IFN-α, or anti PD 1, anti PD L1, anti PD L2, anti CD137, or anti cytotoxic T lymphocyte associated antigen 4 (CTLA 4) antibody (including ipilimumab), or any other antibody or drug specifically targeting T cell co stimulation or immune checkpoint pathways
* Prior therapy with axitinib as well as any prior therapies with other VEGF pathway inhibitors.
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥3), any history of anaphylaxis.
* Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, deep vein thrombosis or symptomatic pulmonary embolism.
* Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines (for example, inactivated influenza vaccines).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2021-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (12):
  - Scottsdale Healthcare Hospitals d/b/a HonorHealth, Scottsdale, Arizona
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Laura & Isaac Perlmutter Cancer Center At NYU Langone, New York, New York
  - NYU Langone Medical Center, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Henry Joyce Cancer Clinic, Nashville, Tennessee
  - University of Utah, Huntsman Cancer Hospital, Salt Lake City, Utah
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
- Japan (3):
  - Niigata University Medical & Dental Hospital, Chuo-ku, Niigata, Niigata
  - Kindai University Hospital, Sayama, Osaka
  - Keio University Hospital, Shinjuku-ku, Tokyo
- United Kingdom (6):
  - Mount Vernon Cancer Center, East and North Herts. NHS Trust, London, Middlesex
  - St Helier Hospital, Carshalton, Surrey
  - St. Bartholomew's Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Rini BI, Atkins MB, Choueiri TK, Teresi RE, Rosbrook B, Thakur M, Hutson TE. Plain language summary looking at how long side effects last after treatment with axitinib is stopped in people with advanced renal cell carcinoma. Future Oncol. 2023 Dec;19(40):2623-2629. doi: 10.2217/fon-2023-0233. Epub 2023 Aug 1. PMID 37526095
- [Derived] Larkin J, Oya M, Martignoni M, Thistlethwaite F, Nathan P, Ornstein MC, Powles T, Beckermann KE, Balar AV, McDermott D, Gupta S, Philips GK, Gordon MS, Uemura H, Tomita Y, Wang J, Michelon E, di Pietro A, Choueiri TK. Avelumab Plus Axitinib as First-Line Therapy for Advanced Renal Cell Carcinoma: Long-Term Results from the JAVELIN Renal 100 Phase Ib Trial. Oncologist. 2023 Apr 6;28(4):333-340. doi: 10.1093/oncolo/oyac243. PMID 36576173
- [Derived] Masters JC, Khandelwal A, di Pietro A, Dai H, Brar S. Model-informed drug development supporting the approval of the avelumab flat-dose regimen in patients with advanced renal cell carcinoma. CPT Pharmacometrics Syst Pharmacol. 2022 Apr;11(4):458-468. doi: 10.1002/psp4.12771. Epub 2022 Feb 27. PMID 35166465
- [Derived] Rini BI, Atkins MB, Choueiri TK, Thomaidou D, Rosbrook B, Thakur M, Hutson TE. Time to Resolution of Axitinib-Related Adverse Events After Treatment Interruption in Patients With Advanced Renal Cell Carcinoma. Clin Genitourin Cancer. 2021 Oct;19(5):e306-e312. doi: 10.1016/j.clgc.2021.03.019. Epub 2021 Apr 5. PMID 33947608
- [Derived] Choueiri TK, Larkin J, Oya M, Thistlethwaite F, Martignoni M, Nathan P, Powles T, McDermott D, Robbins PB, Chism DD, Cho D, Atkins MB, Gordon MS, Gupta S, Uemura H, Tomita Y, Compagnoni A, Fowst C, di Pietro A, Rini BI. Preliminary results for avelumab plus axitinib as first-line therapy in patients with advanced clear-cell renal-cell carcinoma (JAVELIN Renal 100): an open-label, dose-finding and dose-expansion, phase 1b trial. Lancet Oncol. 2018 Apr;19(4):451-460. doi: 10.1016/S1470-2045(18)30107-4. Epub 2018 Mar 9. PMID 29530667
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B9991002&StudyName=A%20Phase%201b%2C%20Open-label%2C%20Dose-finding%20Study%20To%20Evaluate%20Safety%2C%0Apharmacokinetics%20And%20Pharmacodynamics%20Of%20Avelumab%0A%28msb0010718c%29%20In%20Combination%20With%20Axitinib%20%28ag-013736%29%20In%20Patients%0Awith%20Previously%20Untreated%20Advanced%20Renal%20Cell%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, a lead-in period was conducted (only axitinib administered) in few participants prior to the administration of combination treatment (axitinib+avelumab) in treatment period. After 5 years from study initiation, the study was closed by Sponsor due to an internal decision (ie, end of study). No safety concerns were related to the study closure. Data reported based on last participant last visit (LPLV) date (04 March 2021).
Groups:
- Axitinib + Avelumab With Lead-in: Participants received 5 mg axitinib tablets orally twice daily for 7 days in lead-in period (7 days) followed by 10 milligram/ kilogram (mg/kg) avelumab intravenously every 2 weeks along with 5 mg axitinib tablets orally twice daily, on Day 1 of each treatment cycle (duration of each cycle=14 days) in treatment period (up to maximum of 255.4 weeks).
- Axitinib + Avelumab: Participants received 10 mg/kg avelumab intravenously every 2 weeks along with 5 mg axitinib tablets orally twice daily, on Day 1 of each treatment cycle (duration of each cycle=14 days) in treatment period (up to maximum of 240.1 weeks).
Period: Overall Study
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Started | 16 | 39
Completed | 0 | 0
Not Completed | 16 | 39
Not completed — Withdrawal by Subject | 2 | 8
Not completed — Death | 6 | 13
Not completed — Lost to Follow-up | 2 | 3
Not completed — Study closed by Sponsor due to an internal decision with no safety concerns related. | 6 | 15

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab | Total
Number analyzed (Participants) | 16 | 39 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (8.45) | 60.5 (8.89) | 60.3 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 11 | 13
  Male | 14 | 28 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 35 | 51
  Unknown or Not Reported | 0 | 4 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 2 | 3
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 6 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 15 | 29 | 44
  Other | 0 | 1 | 1
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT: greater than or equal to (>=) Grade 3 hematologic/non-hematologic toxicity, Grade 3-4 liver-related laboratory test elevation (alanine aminotransferase, aspartate aminotransferase) with Grade 2 elevation of total bilirubin, non-hematologic Grade 3 laboratory abnormality (required medical intervention to treat participant/led to hospitalization), inability to complete >=75% of first 2 cycles doses of axitinib (from Cycle 1 Day 1 after completion of lead-in period) or 2 infusions of avelumab within DLT observation period due to investigational product related toxicity.
Time Frame: DLT observation period (from the beginning of Cycle 1 up to the end of Cycle 2 [28 days])
Population: DLT evaluable analysis set: First 6 enrolled participants who received at least 1 dose of avelumab and axitinib, and either experienced DLT during DLT observation period or completed it. Data for this endpoint was only planned to be collected and analyzed for "Axitinib + Avelumab with Lead-in" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Avelumab With Lead-in
Number analyzed (Participants) | 6
Participants | 1

2. Secondary Outcome: Number of Participants With All-causality Treatment Emergent Adverse Events (TEAEs)
Description: Adverse event (AE)=any untoward medical occurrence in participant who received study treatment without regard to causality. TEAE=event between first dose of study treatment and up to 30 days after last dose that were absent before treatment or worsened relative to pretreatment state. Serious AE (SAE)=AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience; persistent or significant disability/incapacity; congenital anomaly. AEs were graded by worst National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 severity grade. Grade 3 event=unacceptable or intolerable event, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 event caused participant to be in imminent danger of death. Grade 5 event=death related to AE. The results reflect data available on cutoff of LPLV (04 Mar 2021).
Time Frame: Baseline up to 30 days after the last dose of study treatment (maximum of 259.7 weeks)
Population: The population for this outcome measure included all enrolled participants who received at least 1 dose of avelumab or axitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 16 | 39
Participants
  Participants with TEAEs | 16 | 39
  Participants with Grade >=3 TEAEs | 13 | 30
  Participants with SAEs | 6 | 18

3. Secondary Outcome: Number of Participants With Treatment-related TEAEs
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. TEAE=event between first dose of study treatment and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience; persistent or significant disability/incapacity; congenital anomaly. AEs were graded by worst NCI CTCAE v4.03 severity grade. Grade 3 events=unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 events caused participant to be in imminent danger of death. Grade 5 events=death related to an AE. Treatment-related AEs and SAEs were determined by the investigator. The results reflect data available on cutoff of LPLV (04 Mar 2021).
Time Frame: Baseline up to 30 days after the last dose of study treatment (maximum of 259.7 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 16 | 39
Participants
  Participants with treatment-related TEAEs | 15 | 39
  Participants with Grade >=3 treatment-related TEAEs | 11 | 23
  Participants with treatment-related SAEs | 3 | 10

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities Graded by NCI CTCAE Version 4.03 - Hematology
Description: Laboratory abnormalities (hematology) reported included anemia, platelet count decreased, lymphocyte count decreased, and neutrophil count decreased. Grade 1=mild transient reaction; infusion interruption not indicated; intervention not indicated. Grade 2=therapy or infusion interruption indicated but responds promptly to symptomatic treatment; prophylactic medications indicated for <=24 hours. Grade 3=prolonged; recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae. Grade 4=life threatening consequences; urgent intervention indicated. Grade 5=death. The results reflect data available on cutoff of LPLV (04 Mar 2021).
Time Frame: Baseline up to 30 days after the last dose of study treatment and 1 day before the start day of new anti-cancer drug therapy (maximum of 259.7 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 16 | 39
Participants
  Participants with Grade >=1 anemia | 8 | 24
  Participants with Grade >=3 anemia | 0 | 2
  Participants with Grade >=1 platelet count decreased | 4 | 11
  Participants with Grade >=3 platelet count decreased | 0 | 0
  Participants with Grade >=1 lymphocyte count decreased | 10 | 16
  Participants with Grade >=3 lymphocyte count decreased | 1 | 3
  Participants with Grade >=1 neutrophil count decreased | 1 | 4
  Participants with Grade >=3 neutrophil count decreased | 0 | 0

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities Graded by NCI CTCAE Version 4.03 - Chemistry
Description: Laboratory abnormalities (chemistry) reported included creatinine increased, serum amylase increased, lipase increased, alanine aminotransferase (ALT) increased, aspartate aminotransferase (AST) increased, blood bilirubin increased, creatine kinase increased, hypoglycemia, and hyperglycemia. Grade 1=mild transient reaction; infusion interruption not indicated; intervention not indicated. Grade 2=therapy or infusion interruption indicated but responds promptly to symptomatic treatment; prophylactic medications indicated for <=24 hours. Grade 3=prolonged; recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae. Grade 4=life threatening consequences; urgent intervention indicated. Grade 5=death. The results reflect data available on cutoff of LPLV (04 Mar 2021).
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 16 | 39
Participants
  Participants with Grade >=1 creatinine increased | 16 | 37
  Participants with Grade >=3 creatinine increased | 0 | 0
  Participants with Grade >=1 serum amylase increased | 11 | 16
  Participants with Grade >=3 serum amylase increased | 4 | 3
  Participants with Grade >=1 lipase increased | 9 | 16
  Participants with Grade >=3 lipase increased | 5 | 8
  Participants with Grade >=1 ALT increased | 8 | 20
  Participants with Grade >=3 ALT increased | 2 | 2
  Participants with Grade >=1 AST increased | 10 | 21
  Participants with Grade >=3 AST increased | 1 | 1
  Participants with Grade >=1 blood bilirubin increased | 2 | 7
  Participants with Grade >=3 blood bilirubin increased | 0 | 0
  Participants with Grade >=1 creatine kinase increased | 6 | 15
  Participants with Grade >=3 creatine kinase increased | 1 | 0
  Participants with Grade >=1 hypoglycemia | 4 | 4
  Participants with Grade >=3 hypoglycemia | 0 | 0
  Participants with Grade >=1 hyperglycemia | 5 | 13
  Participants with Grade >=3 hyperglycemia | 2 | 1

6. Secondary Outcome: Change From Baseline in Vital Signs - Sitting Diastolic Blood Pressure
Description: Blood pressure was taken with the participant in the seated position after the participant had been sitting quietly for at least 5 minutes. Baseline was defined as the last assessment prior to the date/time of the first dose of study treatment, which occurred on Day 1 in Lead-in period for participants with lead-in, and occurred on Cycle 1 Day 1 (C1D1) for participants without lead-in. The results reflect data available on cutoff of primary completion date (PCD) (03 Apr 2018).
Time Frame: Baseline, Day 1 of each cycle, Day 8 of Cycles 1 and 2, end of treatment, Follow-up Days 30, 60, 90 for all participants in the analysis population, and Lead-in Day 7 for participants with lead-in (maximum of 139.6 weeks by PCD)
Population: The population for this outcome measure included all enrolled participants who received at least 1 dose of avelumab or axitinib (ie, safety analysis set). Number of Participants Analyzed represents the total number of participants in the safety analysis set. Number Analyzed in each row represents the number of participants in the safety analysis set with at least 1 baseline and 1 post-baseline assessments at the visit.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mm Hg)
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 16 | 39
millimeter of mercury (mm Hg)
  Lead-in Day 7: number analyzed (Participants) | 16 | 0
  Lead-in Day 7 | 5.4 (9.32) |
  C1D1: number analyzed (Participants) | 16 | 0
  C1D1 | 4.1 (9.36) |
  C1D8: number analyzed (Participants) | 12 | 37
  C1D8 | 3.2 (12.80) | 9.8 (11.81)
  C2D1: number analyzed (Participants) | 16 | 38
  C2D1 | 3.4 (13.15) | 10.1 (10.03)
  C2D8: number analyzed (Participants) | 6 | 3
  C2D8 | 1.8 (10.01) | 14.7 (5.03)
  C3D1: number analyzed (Participants) | 14 | 37
  C3D1 | 6.1 (12.16) | 10.2 (11.80)
  C4D1: number analyzed (Participants) | 14 | 37
  C4D1 | 3.6 (10.34) | 8.8 (9.60)
  C5D1: number analyzed (Participants) | 14 | 34
  C5D1 | 4.8 (10.53) | 6.9 (11.64)
  C6D1: number analyzed (Participants) | 14 | 34
  C6D1 | 3.0 (9.84) | 7.5 (11.76)
  C7D1: number analyzed (Participants) | 13 | 33
  C7D1 | 4.8 (11.82) | 7.5 (12.50)
  C8D1: number analyzed (Participants) | 14 | 31
  C8D1 | 5.7 (10.76) | 9.0 (10.86)
  C9D1: number analyzed (Participants) | 14 | 30
  C9D1 | 3.9 (10.80) | 10.0 (13.44)
  C10D1: number analyzed (Participants) | 12 | 29
  C10D1 | 7.3 (9.80) | 7.7 (8.97)
  C11D1: number analyzed (Participants) | 12 | 27
  C11D1 | 7.4 (8.98) | 7.5 (11.09)
  C12D1: number analyzed (Participants) | 12 | 28
  C12D1 | 5.3 (8.20) | 6.6 (12.07)
  C13D1: number analyzed (Participants) | 12 | 27
  C13D1 | 6.0 (7.71) | 10.5 (11.92)
  C14D1: number analyzed (Participants) | 12 | 27
  C14D1 | 5.4 (10.87) | 7.2 (14.04)
  C15D1: number analyzed (Participants) | 12 | 25
  C15D1 | 6.9 (6.56) | 7.6 (12.13)
  C16D1: number analyzed (Participants) | 10 | 24
  C16D1 | 7.5 (10.33) | 5.8 (13.57)
  C17D1: number analyzed (Participants) | 11 | 24
  C17D1 | 6.2 (9.84) | 6.4 (13.20)
  C18D1: number analyzed (Participants) | 11 | 23
  C18D1 | 4.3 (8.45) | 5.1 (12.22)
  C19D1: number analyzed (Participants) | 11 | 22
  C19D1 | 6.3 (7.58) | 5.5 (10.67)
  C20D1: number analyzed (Participants) | 10 | 21
  C20D1 | 7.9 (6.71) | 6.9 (11.69)
  C21D1: number analyzed (Participants) | 10 | 22
  C21D1 | 8.9 (9.35) | 6.6 (10.22)
  C22D1: number analyzed (Participants) | 10 | 19
  C22D1 | 7.2 (9.34) | 6.2 (11.96)
  C23D1: number analyzed (Participants) | 9 | 19
  C23D1 | 9.2 (9.54) | 4.5 (11.52)
  C24D1: number analyzed (Participants) | 10 | 19
  C24D1 | 7.3 (8.42) | 4.3 (12.91)
  C25D1: number analyzed (Participants) | 10 | 20
  C25D1 | 3.1 (9.62) | 6.0 (13.34)
  C26D1: number analyzed (Participants) | 10 | 17
  C26D1 | 5.6 (9.65) | 7.8 (12.33)
  C27D1: number analyzed (Participants) | 10 | 18
  C27D1 | 4.5 (8.64) | 6.2 (13.39)
  C28D1: number analyzed (Participants) | 10 | 18
  C28D1 | 4.9 (7.53) | 6.2 (13.35)
  C29D1: number analyzed (Participants) | 10 | 19
  C29D1 | 5.4 (9.90) | 7.1 (11.13)
  C30D1: number analyzed (Participants) | 10 | 19
  C30D1 | 5.6 (8.53) | 6.1 (13.32)
  C31D1: number analyzed (Participants) | 10 | 18
  C31D1 | 4.8 (11.40) | 6.7 (10.41)
  C32D1: number analyzed (Participants) | 10 | 17
  C32D1 | 7.1 (11.06) | 7.6 (13.52)
  C33D1: number analyzed (Participants) | 10 | 17
  C33D1 | 5.5 (6.59) | 3.6 (13.67)
  C34D1: number analyzed (Participants) | 10 | 17
  C34D1 | 3.5 (13.67) | 5.0 (15.71)
  C35D1: number analyzed (Participants) | 10 | 16
  C35D1 | 7.2 (9.76) | 8.1 (12.46)
  C36D1: number analyzed (Participants) | 10 | 16
  C36D1 | 7.5 (9.40) | 10.9 (11.31)
  C37D1: number analyzed (Participants) | 10 | 16
  C37D1 | 9.9 (10.47) | 7.6 (13.32)
  C38D1: number analyzed (Participants) | 10 | 16
  C38D1 | 5.0 (8.92) | 6.9 (12.73)
  C39D1: number analyzed (Participants) | 9 | 15
  C39D1 | 6.6 (10.10) | 7.9 (14.61)
  C40D1: number analyzed (Participants) | 10 | 16
  C40D1 | 7.8 (10.75) | 6.0 (13.08)
  C41D1: number analyzed (Participants) | 9 | 15
  C41D1 | 6.6 (9.76) | 8.4 (11.70)
  C42D1: number analyzed (Participants) | 9 | 14
  C42D1 | 5.9 (9.35) | 5.7 (13.64)
  C43D1: number analyzed (Participants) | 8 | 13
  C43D1 | 13.0 (11.53) | 2.5 (7.73)
  C44D1: number analyzed (Participants) | 8 | 9
  C44D1 | 8.3 (11.04) | 6.6 (10.08)
  C45D1: number analyzed (Participants) | 8 | 8
  C45D1 | 8.1 (10.23) | 5.4 (13.16)
  C46D1: number analyzed (Participants) | 8 | 8
  C46D1 | 11.1 (11.27) | 3.0 (14.03)
  C47D1: number analyzed (Participants) | 8 | 8
  C47D1 | 8.4 (13.62) | 1.1 (12.01)
  C48D1: number analyzed (Participants) | 8 | 8
  C48D1 | 6.3 (9.75) | 3.9 (13.37)
  C49D1: number analyzed (Participants) | 7 | 8
  C49D1 | 9.4 (10.67) | 11.8 (11.44)
  C50D1: number analyzed (Participants) | 6 | 8
  C50D1 | 9.0 (9.27) | 7.0 (11.53)
  C51D1: number analyzed (Participants) | 6 | 7
  C51D1 | 9.3 (10.17) | 4.3 (10.14)
  C52D1: number analyzed (Participants) | 6 | 5
  C52D1 | 9.3 (11.60) | 8.2 (11.48)
  C53D1: number analyzed (Participants) | 5 | 4
  C53D1 | 15.4 (18.37) | 2.0 (14.72)
  C54D1: number analyzed (Participants) | 4 | 3
  C54D1 | 12.5 (7.42) | 0.3 (12.66)
  C55D1: number analyzed (Participants) | 4 | 1
  C55D1 | 16.0 (19.71) | -3.0 (NA) — Standard deviation was not calculated for n<3.
  C56D1: number analyzed (Participants) | 4 | 1
  C56D1 | 10.0 (13.74) | 0.0 (NA) — Standard deviation was not calculated for n<3.
  C57D1: number analyzed (Participants) | 4 | 0
  C57D1 | 14.5 (12.15) |
  C58D1: number analyzed (Participants) | 4 | 0
  C58D1 | 16.5 (12.82) |
  C59D1: number analyzed (Participants) | 2 | 0
  C59D1 | 26.5 (9.19) |
  C60D1: number analyzed (Participants) | 2 | 0
  C60D1 | 22.5 (4.95) |
  C61D1: number analyzed (Participants) | 2 | 0
  C61D1 | 24.5 (4.95) |
  C62D1: number analyzed (Participants) | 2 | 0
  C62D1 | 22.0 (1.41) |
  End of Treatment: number analyzed (Participants) | 8 | 20
  End of Treatment | -1.6 (10.38) | 2.5 (13.05)
  Follow-up Day 30: number analyzed (Participants) | 5 | 11
  Follow-up Day 30 | -3.2 (8.41) | -2.9 (12.51)
  Follow-up Day 60: number analyzed (Participants) | 3 | 6
  Follow-up Day 60 | -4.7 (10.26) | 3.8 (8.33)
  Follow-up Day 90: number analyzed (Participants) | 3 | 4
  Follow-up Day 90 | -2.0 (4.58) | 1.3 (6.18)

7. Secondary Outcome: Change From Baseline in Vital Signs - Sitting Systolic Blood Pressure
Description: Blood pressure was taken with the participant in the seated position after the participant had been sitting quietly for at least 5 minutes. Baseline was defined as the last assessment prior to the date/time of the first dose of study treatment, which occurred on Day 1 in Lead-in period for participants with lead-in, and occurred on Cycle 1 Day 1 (C1D1) for participants without lead-in. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 16 | 39
mm Hg
  Lead-in Day 7: number analyzed (Participants) | 16 | 0
  Lead-in Day 7 | 9.7 (13.44) |
  C1D1: number analyzed (Participants) | 16 | 0
  C1D1 | 11.0 (18.20) |
  C1D8: number analyzed (Participants) | 12 | 37
  C1D8 | 8.0 (18.94) | 10.3 (16.12)
  C2D1: number analyzed (Participants) | 16 | 38
  C2D1 | 4.6 (18.49) | 11.2 (11.47)
  C2D8: number analyzed (Participants) | 6 | 3
  C2D8 | 0.8 (15.63) | 17.7 (6.66)
  C3D1: number analyzed (Participants) | 14 | 37
  C3D1 | 9.9 (18.96) | 8.7 (15.05)
  C4D1: number analyzed (Participants) | 14 | 37
  C4D1 | 6.7 (15.61) | 5.8 (11.73)
  C5D1: number analyzed (Participants) | 14 | 34
  C5D1 | 6.2 (19.45) | 6.7 (14.90)
  C6D1: number analyzed (Participants) | 14 | 34
  C6D1 | 6.5 (15.05) | 5.2 (13.34)
  C7D1: number analyzed (Participants) | 13 | 33
  C7D1 | 10.2 (14.46) | 6.1 (14.49)
  C8D1: number analyzed (Participants) | 14 | 31
  C8D1 | 13.5 (12.07) | 8.0 (15.14)
  C9D1: number analyzed (Participants) | 14 | 30
  C9D1 | 11.4 (14.24) | 10.2 (16.29)
  C10D1: number analyzed (Participants) | 12 | 29
  C10D1 | 8.9 (16.83) | 8.4 (15.69)
  C11D1: number analyzed (Participants) | 12 | 27
  C11D1 | 7.8 (15.36) | 7.2 (14.83)
  C12D1: number analyzed (Participants) | 12 | 28
  C12D1 | 6.8 (11.27) | 4.1 (14.29)
  C13D1: number analyzed (Participants) | 12 | 27
  C13D1 | 7.3 (11.17) | 8.6 (16.01)
  C14D1: number analyzed (Participants) | 12 | 27
  C14D1 | 5.8 (15.49) | 3.9 (17.66)
  C15D1: number analyzed (Participants) | 12 | 25
  C15D1 | 7.3 (13.89) | 7.3 (20.46)
  C16D1: number analyzed (Participants) | 10 | 24
  C16D1 | 6.2 (13.46) | 5.5 (16.80)
  C17D1: number analyzed (Participants) | 11 | 24
  C17D1 | 7.3 (15.55) | 3.5 (17.32)
  C18D1: number analyzed (Participants) | 11 | 23
  C18D1 | 3.5 (14.67) | 4.2 (15.07)
  C19D1: number analyzed (Participants) | 11 | 22
  C19D1 | 5.8 (16.04) | 2.6 (14.15)
  C20D1: number analyzed (Participants) | 10 | 21
  C20D1 | 8.3 (9.67) | 1.1 (12.20)
  C21D1: number analyzed (Participants) | 10 | 22
  C21D1 | 5.0 (14.14) | 3.1 (10.17)
  C22D1: number analyzed (Participants) | 10 | 19
  C22D1 | 2.9 (14.53) | 0.2 (14.31)
  C23D1: number analyzed (Participants) | 9 | 19
  C23D1 | 9.3 (14.19) | 1.5 (15.05)
  C24D1: number analyzed (Participants) | 10 | 19
  C24D1 | 9.1 (12.55) | -0.1 (16.57)
  C25D1: number analyzed (Participants) | 10 | 20
  C25D1 | 4.0 (12.78) | 3.5 (15.28)
  C26D1: number analyzed (Participants) | 10 | 17
  C26D1 | 2.8 (15.86) | 3.4 (15.82)
  C27D1: number analyzed (Participants) | 10 | 18
  C27D1 | 5.4 (14.74) | 1.6 (16.13)
  C28D1: number analyzed (Participants) | 10 | 18
  C28D1 | 7.8 (14.49) | 2.1 (16.65)
  C29D1: number analyzed (Participants) | 10 | 19
  C29D1 | 3.3 (14.28) | 4.1 (11.82)
  C30D1: number analyzed (Participants) | 10 | 19
  C30D1 | 6.4 (13.57) | 2.9 (15.17)
  C31D1: number analyzed (Participants) | 10 | 18
  C31D1 | 2.7 (13.14) | 1.7 (10.52)
  C32D1: number analyzed (Participants) | 10 | 17
  C32D1 | 8.6 (16.71) | 3.8 (14.22)
  C33D1: number analyzed (Participants) | 10 | 17
  C33D1 | 2.9 (16.07) | 0.2 (15.02)
  C34D1: number analyzed (Participants) | 10 | 17
  C34D1 | 2.8 (18.79) | 2.5 (15.97)
  C35D1: number analyzed (Participants) | 10 | 16
  C35D1 | 10.3 (13.47) | 2.9 (12.89)
  C36D1: number analyzed (Participants) | 10 | 16
  C36D1 | 9.0 (12.92) | 5.3 (19.01)
  C37D1: number analyzed (Participants) | 10 | 16
  C37D1 | 10.2 (11.48) | 2.7 (16.02)
  C38D1: number analyzed (Participants) | 10 | 16
  C38D1 | 8.3 (11.83) | 4.9 (14.66)
  C39D1: number analyzed (Participants) | 9 | 15
  C39D1 | 3.8 (13.33) | 4.3 (15.83)
  C40D1: number analyzed (Participants) | 10 | 16
  C40D1 | 10.9 (14.13) | 3.8 (12.86)
  C41D1: number analyzed (Participants) | 9 | 15
  C41D1 | 7.9 (16.74) | 3.7 (14.22)
  C42D1: number analyzed (Participants) | 9 | 14
  C42D1 | 11.6 (15.74) | 0.9 (15.02)
  C43D1: number analyzed (Participants) | 8 | 13
  C43D1 | 12.3 (13.20) | -1.9 (11.49)
  C44D1: number analyzed (Participants) | 8 | 9
  C44D1 | 9.6 (21.41) | 0.8 (5.70)
  C45D1: number analyzed (Participants) | 8 | 8
  C45D1 | 9.1 (17.71) | -3.5 (14.18)
  C46D1: number analyzed (Participants) | 8 | 8
  C46D1 | 6.1 (11.28) | -3.4 (10.65)
  C47D1: number analyzed (Participants) | 8 | 8
  C47D1 | 6.6 (18.31) | 2.8 (13.29)
  C48D1: number analyzed (Participants) | 8 | 8
  C48D1 | -0.1 (15.04) | -1.3 (9.50)
  C49D1: number analyzed (Participants) | 7 | 8
  C49D1 | 5.4 (13.73) | 7.0 (14.11)
  C50D1: number analyzed (Participants) | 6 | 8
  C50D1 | 9.7 (10.50) | 0.9 (10.06)
  C51D1: number analyzed (Participants) | 6 | 7
  C51D1 | 13.5 (13.85) | 1.4 (10.01)
  C52D1: number analyzed (Participants) | 6 | 5
  C52D1 | 4.3 (16.17) | 5.4 (17.74)
  C53D1: number analyzed (Participants) | 5 | 4
  C53D1 | 17.0 (16.29) | 1.5 (17.94)
  C54D1: number analyzed (Participants) | 4 | 3
  C54D1 | 10.8 (14.20) | 0.0 (18.36)
  C55D1: number analyzed (Participants) | 4 | 1
  C55D1 | 15.8 (19.17) | 6.0 (NA) — Standard deviation was not calculated for n<3.
  C56D1: number analyzed (Participants) | 4 | 1
  C56D1 | 8.5 (11.62) | 3.0 (NA) — Standard deviation was not calculated for n<3.
  C57D1: number analyzed (Participants) | 4 | 0
  C57D1 | 11.5 (12.23) |
  C58D1: number analyzed (Participants) | 4 | 0
  C58D1 | 8.0 (17.45) |
  C59D1: number analyzed (Participants) | 2 | 0
  C59D1 | 21.5 (4.95) |
  C60D1: number analyzed (Participants) | 2 | 0
  C60D1 | 22.0 (19.80) |
  C61D1: number analyzed (Participants) | 2 | 0
  C61D1 | 20.0 (15.56) |
  C62D1: number analyzed (Participants) | 2 | 0
  C62D1 | 14.5 (13.44) |
  End of Treatment: number analyzed (Participants) | 8 | 20
  End of Treatment | 11.3 (25.45) | 3.5 (18.94)
  Follow-up Day 30: number analyzed (Participants) | 5 | 11
  Follow-up Day 30 | 15.0 (20.65) | 1.7 (18.67)
  Follow-up Day 60: number analyzed (Participants) | 3 | 6
  Follow-up Day 60 | 16.0 (9.54) | 15.3 (15.68)
  Follow-up Day 90: number analyzed (Participants) | 3 | 4
  Follow-up Day 90 | 20.7 (13.32) | 9.3 (10.24)

8. Secondary Outcome: Change From Baseline in Vital Signs - Pulse Rate
Description: Pulse rate was taken with the participant in the seated position after the participant had been sitting quietly for at least 5 minutes. Baseline was defined as the last assessment prior to the date/time of the first dose of study treatment, which occurred on Day 1 in Lead-in period for participants with lead-in, and occurred on Cycle 1 Day 1 (C1D1) for participants without lead-in. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: beats per minute (bpm)
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 16 | 39
beats per minute (bpm)
  Lean-in Day 7: number analyzed (Participants) | 16 | 0
  Lean-in Day 7 | -0.5 [-16.0 to 28.0] |
  C1D1: number analyzed (Participants) | 16 | 0
  C1D1 | -1.0 [-21.0 to 19.0] |
  C1D8: number analyzed (Participants) | 12 | 37
  C1D8 | -2.0 [-20.0 to 24.0] | -2.0 [-27.0 to 41.0]
  C2D1: number analyzed (Participants) | 16 | 38
  C2D1 | 3.0 [-20.0 to 24.0] | 4.0 [-30.0 to 29.0]
  C2D8: number analyzed (Participants) | 6 | 3
  C2D8 | 8.0 [-6.0 to 25.0] | 2.0 [-14.0 to 10.0]
  C3D1: number analyzed (Participants) | 14 | 37
  C3D1 | 4.0 [-25.0 to 29.0] | 2.0 [-34.0 to 35.0]
  C4D1: number analyzed (Participants) | 14 | 37
  C4D1 | 1.5 [-20.0 to 24.0] | 4.0 [-28.0 to 48.0]
  C5D1: number analyzed (Participants) | 14 | 34
  C5D1 | 0.0 [-27.0 to 16.0] | 2.5 [-40.0 to 26.0]
  C6D1: number analyzed (Participants) | 14 | 34
  C6D1 | -3.5 [-27.0 to 35.0] | 3.5 [-32.0 to 35.0]
  C7D1: number analyzed (Participants) | 13 | 33
  C7D1 | 1.0 [-26.0 to 20.0] | 1.0 [-42.0 to 34.0]
  C8D1: number analyzed (Participants) | 14 | 31
  C8D1 | -6.5 [-34.0 to 13.0] | -1.0 [-40.0 to 46.0]
  C9D1: number analyzed (Participants) | 14 | 30
  C9D1 | -1.5 [-26.0 to 25.0] | 1.0 [-35.0 to 30.0]
  C10D1: number analyzed (Participants) | 12 | 29
  C10D1 | -3.0 [-33.0 to 17.0] | 3.0 [-34.0 to 43.0]
  C11D1: number analyzed (Participants) | 12 | 27
  C11D1 | -2.0 [-30.0 to 22.0] | 3.0 [-37.0 to 41.0]
  C12D1: number analyzed (Participants) | 12 | 28
  C12D1 | -6.0 [-33.0 to 5.0] | 1.5 [-23.0 to 33.0]
  C13D1: number analyzed (Participants) | 12 | 27
  C13D1 | -1.5 [-33.0 to 25.0] | 2.0 [-28.0 to 44.0]
  C14D1: number analyzed (Participants) | 12 | 27
  C14D1 | 1.5 [-32.0 to 29.0] | 5.0 [-37.0 to 45.0]
  C15D1: number analyzed (Participants) | 12 | 25
  C15D1 | -4.5 [-31.0 to 42.0] | -3.0 [-31.0 to 32.0]
  C16D1: number analyzed (Participants) | 10 | 24
  C16D1 | -1.0 [-18.0 to 30.0] | 1.5 [-36.0 to 40.0]
  C17D1: number analyzed (Participants) | 11 | 24
  C17D1 | -6.0 [-38.0 to 32.0] | 1.5 [-32.0 to 41.0]
  C18D1: number analyzed (Participants) | 11 | 23
  C18D1 | 0.0 [-30.0 to 21.0] | 3.0 [-37.0 to 41.0]
  C19D1: number analyzed (Participants) | 11 | 22
  C19D1 | -1.0 [-28.0 to 29.0] | -3.0 [-43.0 to 22.0]
  C20D1: number analyzed (Participants) | 10 | 21
  C20D1 | 2.0 [-30.0 to 26.0] | 1.0 [-35.0 to 24.0]
  C21D1: number analyzed (Participants) | 10 | 22
  C21D1 | -1.5 [-21.0 to 24.0] | 2.5 [-31.0 to 59.0]
  C22D1: number analyzed (Participants) | 10 | 19
  C22D1 | 0.0 [-12.0 to 27.0] | -6.0 [-33.0 to 20.0]
  C23D1: number analyzed (Participants) | 9 | 19
  C23D1 | 2.0 [-20.0 to 17.0] | -3.0 [-33.0 to 24.0]
  C24D1: number analyzed (Participants) | 10 | 19
  C24D1 | -3.5 [-25.0 to 12.0] | 0.0 [-30.0 to 25.0]
  C25D1: number analyzed (Participants) | 10 | 20
  C25D1 | 0.0 [-15.0 to 16.0] | -4.5 [-29.0 to 18.0]
  C26D1: number analyzed (Participants) | 10 | 17
  C26D1 | -4.0 [-25.0 to 17.0] | -3.0 [-30.0 to 19.0]
  C27D1: number analyzed (Participants) | 10 | 18
  C27D1 | 1.5 [-11.0 to 11.0] | 0.5 [-28.0 to 19.0]
  C28D1: number analyzed (Participants) | 10 | 18
  C28D1 | -8.5 [-21.0 to 9.0] | 0.5 [-29.0 to 34.0]
  C29D1: number analyzed (Participants) | 10 | 19
  C29D1 | -6.0 [-17.0 to 12.0] | -4.0 [-31.0 to 22.0]
  C30D1: number analyzed (Participants) | 10 | 19
  C30D1 | -3.0 [-16.0 to 17.0] | -2.0 [-26.0 to 17.0]
  C31D1: number analyzed (Participants) | 10 | 18
  C31D1 | 1.5 [-22.0 to 11.0] | -3.5 [-20.0 to 24.0]
  C32D1: number analyzed (Participants) | 10 | 17
  C32D1 | 2.0 [-22.0 to 12.0] | 2.0 [-32.0 to 38.0]
  C33D1: number analyzed (Participants) | 10 | 17
  C33D1 | -4.0 [-26.0 to 13.0] | 1.0 [-25.0 to 14.0]
  C34D1: number analyzed (Participants) | 10 | 17
  C34D1 | -1.0 [-25.0 to 38.0] | 1.0 [-19.0 to 14.0]
  C35D1: number analyzed (Participants) | 10 | 16
  C35D1 | -2.0 [-27.0 to 21.0] | 2.5 [-19.0 to 27.0]
  C36D1: number analyzed (Participants) | 10 | 16
  C36D1 | 1.0 [-20.0 to 14.0] | 0.0 [-19.0 to 28.0]
  C37D1: number analyzed (Participants) | 10 | 16
  C37D1 | 1.5 [-26.0 to 19.0] | 0.0 [-14.0 to 24.0]
  C38D1: number analyzed (Participants) | 10 | 16
  C38D1 | -1.0 [-24.0 to 26.0] | 2.0 [-16.0 to 24.0]
  C39D1: number analyzed (Participants) | 9 | 15
  C39D1 | 0.0 [-24.0 to 12.0] | -1.0 [-13.0 to 23.0]
  C40D1: number analyzed (Participants) | 10 | 16
  C40D1 | -3.0 [-29.0 to 24.0] | 2.5 [-18.0 to 25.0]
  C41D1: number analyzed (Participants) | 9 | 15
  C41D1 | -5.0 [-28.0 to 21.0] | 1.0 [-18.0 to 17.0]
  C42D1: number analyzed (Participants) | 9 | 14
  C42D1 | -3.0 [-24.0 to 12.0] | 0.0 [-17.0 to 14.0]
  C43D1: number analyzed (Participants) | 8 | 13
  C43D1 | 4.5 [-16.0 to 12.0] | 1.0 [-19.0 to 20.0]
  C44D1: number analyzed (Participants) | 8 | 9
  C44D1 | 2.0 [-13.0 to 19.0] | 5.0 [-7.0 to 29.0]
  C45D1: number analyzed (Participants) | 8 | 8
  C45D1 | 2.5 [-12.0 to 18.0] | 9.5 [-8.0 to 18.0]
  C46D1: number analyzed (Participants) | 8 | 8
  C46D1 | 1.0 [-16.0 to 25.0] | 11.5 [-4.0 to 22.0]
  C47D1: number analyzed (Participants) | 8 | 8
  C47D1 | 5.0 [-7.0 to 35.0] | 5.5 [-5.0 to 24.0]
  C48D1: number analyzed (Participants) | 8 | 8
  C48D1 | -3.0 [-20.0 to 29.0] | 4.5 [-13.0 to 16.0]
  C49D1: number analyzed (Participants) | 7 | 8
  C49D1 | 10.0 [-14.0 to 23.0] | -0.5 [-12.0 to 13.0]
  C50D1: number analyzed (Participants) | 6 | 8
  C50D1 | -2.0 [-14.0 to 11.0] | 4.0 [-16.0 to 15.0]
  C51D1: number analyzed (Participants) | 6 | 7
  C51D1 | 0.0 [-8.0 to 11.0] | 6.0 [-4.0 to 14.0]
  C52D1: number analyzed (Participants) | 6 | 5
  C52D1 | 0.5 [-12.0 to 12.0] | 3.0 [-6.0 to 20.0]
  C53D1: number analyzed (Participants) | 5 | 4
  C53D1 | 6.0 [-14.0 to 11.0] | 10.0 [-3.0 to 17.0]
  C54D1: number analyzed (Participants) | 4 | 3
  C54D1 | 2.5 [-6.0 to 6.0] | 1.0 [-2.0 to 4.0]
  C55D1: number analyzed (Participants) | 4 | 1
  C55D1 | -6.5 [-9.0 to 7.0] | 5.0 [5.0 to 5.0]
  C56D1: number analyzed (Participants) | 4 | 1
  C56D1 | 1.5 [-10.0 to 10.0] | 1.0 [1.0 to 1.0]
  C57D1: number analyzed (Participants) | 4 | 0
  C57D1 | -4.0 [-17.0 to 6.0] |
  C58D1: number analyzed (Participants) | 4 | 0
  C58D1 | 4.0 [-15.0 to 9.0] |
  C59D1: number analyzed (Participants) | 2 | 0
  C59D1 | 2.0 [-7.0 to 11.0] |
  C60D1: number analyzed (Participants) | 2 | 0
  C60D1 | 1.5 [-11.0 to 14.0] |
  C61D1: number analyzed (Participants) | 2 | 0
  C61D1 | 2.0 [-8.0 to 12.0] |
  C62D1: number analyzed (Participants) | 2 | 0
  C62D1 | 9.0 [-1.0 to 19.0] |
  End of Treatment: number analyzed (Participants) | 8 | 20
  End of Treatment | 2.5 [-32.0 to 9.0] | 6.5 [-25.0 to 44.0]
  Follow-up Day 30: number analyzed (Participants) | 5 | 11
  Follow-up Day 30 | -1.0 [-26.0 to 2.0] | -2.0 [-38.0 to 51.0]
  Follow-up Day 60: number analyzed (Participants) | 3 | 6
  Follow-up Day 60 | 2.0 [-23.0 to 29.0] | 3.0 [-11.0 to 43.0]
  Follow-up Day 90: number analyzed (Participants) | 3 | 4
  Follow-up Day 90 | 9.0 [-23.0 to 11.0] | 5.5 [-7.0 to 50.0]

9. Secondary Outcome: Number of Participants Achieving Objective Response (OR) Based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Confirmed OR was defined as complete response (CR) or partial response (PR) according to RECIST v1.1 from the start date until disease progression or death due to any cause. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR was defined as >= 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. All target lesions must have been assessed. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Cycle 1 Day 1 up to 30 months after the first dose
Population: The population for this outcome measure included all participants who received at least 1 dose of study drug (axitinib or avelumab) and all participants who were randomized independent of whether they had received a dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 16 | 39
Participants
  CR | 2 | 2
  PR | 8 | 21

10. Secondary Outcome: Number of Participants Achieving Disease Control (DC) Based on RECIST Version 1.1
Description: DC was defined as OR (CR or PR) or stable disease (SD) per RECIST v1.1 from the start date until the first documentation of objective disease progression or death due to any cause. SD was defined as not qualifying for CR, PR, or progression (PD). PD was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR was defined as >= 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. All target lesions must have been assessed. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Cycle 1 Day 1 up to 30 months after the first dose
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 16 | 39
Participants | 15 | 28

11. Secondary Outcome: Duration of Response (DR) Based on RECIST Version 1.1
Description: DR was defined as the time from the first documentation of objective tumor response (CR or PR) that was subsequently confirmed to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR was defined as >= 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. All target lesions must have been assessed. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Cycle 1 Day 1 up to 30 months after the first dose
Population: The population for this outcome measure included all participants who received at least 1 dose of study drug (axitinib or avelumab), all participants who were randomized independent of whether they had received a dose of study drug, and all participants who had achieved confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 10 | 23
months | NA [4.2 to NA] — Median and upper limit were not estimable. The median DR based on the Kaplan-Meier method had not been reached at the time of data cutoff (03 April 2018). | NA [9.6 to NA] — Median and upper limit were not estimable. The median DR based on the Kaplan-Meier method had not been reached at the time of data cutoff (03 April 2018).

12. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as defined as the time from the start date to the date of the first documentation of objective progression of disease (PD) or death due to any cause, whichever occurred first. PD was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm. All target lesions must have been assessed. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Cycle 1 Day 1 up to 30 months after the first dose
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 16 | 39
months | 19.2 [4.4 to NA] — Upper limit was not estimable. The upper limit for PFS based on the Kaplan-Meier method had not been reached at the time of data cutoff (03 April 2018). | 7.6 [4.1 to NA] — Upper limit was not estimable. The upper limit for PFS based on the Kaplan-Meier method had not been reached at the time of data cutoff (03 April 2018).

13. Secondary Outcome: Time to Tumor Response (TTR) Based on RECIST Version 1.1
Description: TTR was defined as the time from start date to the first documentation of objective tumor response (CR or PR) that was subsequently confirmed. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR was defined as >= 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. All target lesions must have been assessed. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Cycle 1 Day 1 up to 30 months after the first dose
Population: as for outcome 11
Measure: Median (Full Range); unit: months
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 10 | 23
months | 1.6 [1.3 to 5.8] | 1.4 [1.2 to 9.6]

14. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the start date to the date of death due to any cause. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Cycle 1 Day 1 up to 30 months after the first dose
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 16 | 39
months | NA [23.0 to NA] — Median and upper limit were not estimable. The median and upper limit for OS based on the Kaplan-Meier method had not been reached at the time of data cutoff (03 April 2018). | NA [20.1 to NA] — Median and upper limit were not estimable. The median and upper limit for OS based on the Kaplan-Meier method had not been reached at the time of data cutoff (03 April 2018).

15. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Axitinib When Dosed Alone and in Combination With Avelumab
Description: Cmax for axitinib when dosed alone on Lead-in Day 7 and in combination with avelumab on Cycle 4 Day 1 for Axitinib + Avelumab with Lead-in Arm. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Predose, 1, 2, 3, 4, 6, and 8 hours post dose on Lead-in Day 7 and Cycle 4 Day 1
Population: The population for this outcome measure included all enrolled participants who received at least 1 dose of avelumab or axitinib and who had at least 1 of the pharmacokinetic (PK) parameters of interest of either study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Axitinib + Avelumab With Lead-in
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL)
  Lean-in Day 7 | 23.1947 (178)
  Cycle 4 Day 1 | 16.5806 (254)

16. Secondary Outcome: Time for Cmax (Tmax) for Axitinib When Dosed Alone and in Combination With Avelumab
Description: Tmax for axitinib when dosed alone on Lead-in Day 7 and in combination with avelumab on Cycle 4 Day 1 for Axitinib + Avelumab with Lead-in Arm. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Predose, 1, 2, 3, 4, 6, and 8 hours post dose on Lead-in Day 7 and Cycle 4 Day 1
Population: as for outcome 15
Measure: Median (Full Range); unit: hours (hrs)
Arm/Group | Axitinib + Avelumab With Lead-in
Number analyzed (Participants) | 14
hours (hrs)
  Lean-in Day 7 | 2.0900 [0.0170 to 4.1800]
  Cycle 4 Day 1 | 1.9850 [1.0000 to 3.0200]

17. Secondary Outcome: Area Under the Plasma Concentration Time Profile From Time Zero to the Next Dose at Steady State (AUCtau) for Axitinib When Dosed Alone and in Combination With Avelumab
Description: AUCtau was defined as area under the plasma concentration time profile from time zero to time tau, the dosing interval at steady state. tau = 12 hrs for Axitinib. AUCtau for Axitinib when dosed alone on Lead-in Day 7 and in combination with avelumab on Cycle 4 Day 1 for Axitinib + Avelumab with Lead-in Arm was reported. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Predose, 1, 2, 3, 4, 6, and 8 hours post dose on Lead-in Day 7 and Cycle 4 Day 1
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/mL)
Arm/Group | Axitinib + Avelumab With Lead-in
Number analyzed (Participants) | 13
nanograms*hour/milliliter (ng*hr/mL)
  Lean-in Day 7 | 113.11 (206)
  Cycle 4 Day 1 | 95.60 (162)

18. Secondary Outcome: Terminal Half-Life (t1/2) for Axitinib When Dosed Alone and in Combination With Avelumab
Description: t1/2 was calculated by Log e(2)/kel. kel was the terminal phase rate constant calculated by a linear regression of the log linear concentration time-curve. Only those data points judged to describe the terminal log linear decline were used in the regression. t1/2 for Axitinib when dosed alone on Lead-in Day 7 and in combination with avelumab on Cycle 4 Day 1 for Axitinib + Avelumab with Lead-in Arm was reported. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Predose, 1, 2, 3, 4, 6, and 8 hours post dose on Lead-in Day 7 and Cycle 4 Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Axitinib + Avelumab With Lead-in
Number analyzed (Participants) | 10
hrs
  Lean-in Day 7 | 2.755 (1.5417)
  Cycle 4 Day 1 | 3.252 (1.3389)

19. Secondary Outcome: Predose Concentration During Multiple Dosing (Ctrough) for Avelumab
Description: Ctrough was directly observed from data. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Predose on Day 1 of Cycles 1, 2, 3, 4, 6, 8, 14, 20, 26, 32, 38, 44, and 50
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (ug/mL)
Groups:
- All Participants: Participants received 10 mg/kg avelumab intravenously every 2 weeks along with 5 mg axitinib tablets orally twice daily, on Day 1 of each treatment cycle (duration of each cycle=14 days) in treatment period (up to maximum of 255.4 weeks).
Arm/Group | All Participants
Number analyzed (Participants) | 54
microgram per milliliter (ug/mL)
  Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 50
  Cycle 1 Day 1 (C1D1) | 1.0 (181)
  C2D1: number analyzed (Participants) | 51
  C2D1 | 20.3 (82)
  C3D1: number analyzed (Participants) | 32
  C3D1 | 23.9 (151)
  C4D1: number analyzed (Participants) | 36
  C4D1 | 23.4 (103)
  C6D1: number analyzed (Participants) | 31
  C6D1 | 26.3 (134)
  C8D1: number analyzed (Participants) | 30
  C8D1 | 28.3 (106)
  C14D1: number analyzed (Participants) | 28
  C14D1 | 36.1 (59)
  C20D1: number analyzed (Participants) | 21
  C20D1 | 41.0 (60)
  C26D1: number analyzed (Participants) | 14
  C26D1 | 38.4 (77)
  C32D1: number analyzed (Participants) | 14
  C32D1 | 40.8 (72)
  C38D1: number analyzed (Participants) | 13
  C38D1 | 44.5 (68)
  C44D1: number analyzed (Participants) | 4
  C44D1 | 67.5 (52)
  C50D1: number analyzed (Participants) | 2
  C50D1 | 40.5 (121)

20. Secondary Outcome: Cmax for Avelumab
Description: Cmax for avelumab on Cycle 1 Day (C1D1) and C1D4 were reported. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Predose, 1 hour, and 168 hours post dose on Cycle 1 Day 1; predose and 1 hour post dose on Cycle 4 Day 1
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | All Participants
Number analyzed (Participants) | 54
ug/mL
  C1D1: number analyzed (Participants) | 50
  C1D1 | 233.4 (27)
  C4D1: number analyzed (Participants) | 40
  C4D1 | 278.0 (60)

21. Secondary Outcome: Number of Participants With Their Target Programmed Death-Ligand (PD-L1) Status at Baseline
Description: Number of participants with PD-L1 positive (PD-L1 >=1%) status in immune cell (IC), tumor cell (TC), or both IC and TC. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Baseline
Population: The population for this outcome measure included all enrolled participants who had at least 1 screening biomarker assessment and who received at least 1 dose of avelumab or axitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 16 | 39
Participants
  IC | 11 | 30
  TC | 3 | 15
  IC+TC | 11 | 32

22. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADA) Against Avelumab When Combined With Axitinib by Never and Ever Positive Status
Description: Whole blood specimens were collected at the designated times (Day 1 of Cycles 1-4, 6, and 8, then every 12 weeks until Cycle 50, and Follow-up Day 30) to provide serum for evaluation of avelumab immunogenicity. Human serum ADA specimens were analyzed for the presence or absence of anti-avelumab antibodies with quasi-quantitative enzyme-linked immunosorbent assay, following a tiered approach using screening, confirmation and titer/quantitation. ADA serum specimens were screened at tier 1. In the event that there were no positive specimens, no further analyses were to be conducted. If positive specimens were identified, these specimens were further tested with the confirmatory assay to confirm as positive. Number of participants with ADA positive at baseline, ADA never-positive, ADA ever-positive, treatment-boosted ADA, treatment-induced ADA, transient ADA response, or persistent ADA response from baseline up to 2 years. The results reflect data available on cutoff of PCD (03 Apr 2018).
Time Frame: Pre-dose on Day 1 of Cycles 1-4, 6, 8, then every 12 weeks thereafter until Cycle 50, and on Follow-up Day 30 (maximum of 2 years)
Population: The analysis population (ie, Number of Participants Analyzed)=number of participants (#p) received at least 1 dose of study drug and with at least 1 ADA sample collected. Number Analyzed =Number of Participants Analyzed for ADA_p and ADA_n; = #p with valid baseline ADA result for ADA_bp; = #p with valid baseline and at least 1 valid post-baseline ADA results for Tb_ADA; = #p with at least 1 valid post-baseline ADA result and without positive baseline ADA result for Ti_ADA, t_ADA, and p_ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
Number analyzed (Participants) | 15 | 39
Participants
  ADA positive at baseline (ADA_bp): number analyzed (Participants) | 15 | 36
  ADA positive at baseline (ADA_bp) | 2 | 0
  ADA never-positive (ADA_n) | 12 | 31
  ADA ever-positive (ADA_p) | 3 | 8
  Treatment-boosted ADA (Tb_ADA): number analyzed (Participants) | 15 | 35
  Treatment-boosted ADA (Tb_ADA) | 0 | 0
  Treatment-induced ADA (Ti_ADA): number analyzed (Participants) | 13 | 38
  Treatment-induced ADA (Ti_ADA) | 1 | 8
  Transient ADA response (t_ADA): number analyzed (Participants) | 13 | 38
  Transient ADA response (t_ADA) | 0 | 5
  Persistent ADA response (p_ADA): number analyzed (Participants) | 13 | 38
  Persistent ADA response (p_ADA) | 1 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study treatment (maximum duration of 259.7 weeks for participants with Lead-in, and maximum duration of 244.4 weeks for participants without lead-in)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Axitinib + Avelumab With Lead-in | Axitinib + Avelumab
All-Cause Mortality (participants affected / at risk) | 6/16 | 14/39
Serious Adverse Events (participants affected / at risk) | 6/16 | 18/39
Other Adverse Events (participants affected / at risk) | 16/16 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Avelumab With Lead-in (N=16) | Axitinib + Avelumab (N=39)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Amylase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 2
Spinal cord compression (Nervous system disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 2
Haemorrhage (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Avelumab With Lead-in (N=16) | Axitinib + Avelumab (N=39)
Anaemia (Blood and lymphatic system disorders) | 2 | 5
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 2
Hypoacusis (Ear and labyrinth disorders) | 2 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 3
Hypothyroidism (Endocrine disorders) | 4 | 11
Dry eye (Eye disorders) | 1 | 3
Eye haemorrhage (Eye disorders) | 1 | 0
Eyelid irritation (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Anal haemorrhage (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 8 | 12
Dental caries (Gastrointestinal disorders) | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 13 | 26
Diverticulum (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Flatulence (Gastrointestinal disorders) | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 5
Gingival hypertrophy (Gastrointestinal disorders) | 1 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 7 | 8
Oral pain (Gastrointestinal disorders) | 1 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 4 | 4
Tongue discomfort (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 4 | 10
Axillary pain (General disorders) | 0 | 2
Chest discomfort (General disorders) | 2 | 1
Chest pain (General disorders) | 2 | 0
Chills (General disorders) | 2 | 7
Fatigue (General disorders) | 10 | 20
Feeling abnormal (General disorders) | 1 | 0
Feeling cold (General disorders) | 1 | 1
Gait disturbance (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 2
Mucosal inflammation (General disorders) | 2 | 11
Oedema (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 2 | 6
Pain (General disorders) | 1 | 4
Peripheral swelling (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 5
Cellulitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 4 | 5
Rhinitis (Infections and infestations) | 0 | 3
Sinusitis (Infections and infestations) | 1 | 2
Tooth infection (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 7
Urinary tract infection (Infections and infestations) | 2 | 5
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 8
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 6 | 12
Amylase increased (Investigations) | 9 | 10
Aspartate aminotransferase increased (Investigations) | 4 | 14
Blood alkaline phosphatase increased (Investigations) | 1 | 6
Blood bilirubin increased (Investigations) | 1 | 2
Blood cholesterol increased (Investigations) | 2 | 3
Blood corticotrophin decreased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 3
Blood creatinine increased (Investigations) | 5 | 4
Blood lactate dehydrogenase increased (Investigations) | 1 | 1
Blood magnesium decreased (Investigations) | 2 | 0
Blood phosphorus decreased (Investigations) | 3 | 0
Blood sodium decreased (Investigations) | 2 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 1
Blood thyroid stimulating hormone increased (Investigations) | 2 | 1
Blood triglycerides increased (Investigations) | 0 | 3
Blood uric acid increased (Investigations) | 1 | 1
C-reactive protein increased (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 3 | 4
Haemoglobin increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 6 | 7
Lymphocyte count decreased (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 2 | 4
Weight decreased (Investigations) | 2 | 9
Weight increased (Investigations) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 3 | 10
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Gout (Metabolism and nutrition disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Ataxia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 4
Dysgeusia (Nervous system disorders) | 1 | 6
Headache (Nervous system disorders) | 7 | 8
Hyperaesthesia (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 3 | 1
Paraesthesia (Nervous system disorders) | 2 | 3
Tremor (Nervous system disorders) | 2 | 1
Confusional state (Psychiatric disorders) | 1 | 2
Dysphoria (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 6
Mood altered (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 3 | 6
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Balanoposthitis (Reproductive system and breast disorders) | 2 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 4
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 10
Rash (Skin and subcutaneous tissue disorders) | 6 | 15
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 8 | 19
Hypotension (Vascular disorders) | 1 | 5
Ear congestion (Ear and labyrinth disorders) | 1 | 0
Blepharitis (Eye disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Hyperaesthesia teeth (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Multiple allergies (Immune system disorders) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 1
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Blood corticotrophin increased (Investigations) | 0 | 2
White blood cell count decreased (Investigations) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 3
Neurotoxicity (Nervous system disorders) | 1 | 0
Taste disorder (Nervous system disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3
Scar pain (Skin and subcutaneous tissue disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Defaecation urgency (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT02493751/Prot_001.pdf
  • Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT02493751/SAP_000.pdf